CLINICAL TRIAL: NCT04375878
Title: OPTION 2: A Phase 2, Open-Label, Multicenter, 2x2 Crossover Trial to Assess the Safety and Efficacy of MS1819 in Enteric Capsules in Patients With Exocrine Pancreatic Insufficiency Due to Cystic Fibrosis; With an Extension Phase Evaluation of Immediate Release MS1819 Capsules
Brief Title: OPTION 2: A Trial to Assess the Safety and Efficacy of MS1819 in Enteric Capsules in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Entero Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AZ-CF2002
Record Dates: First submitted 2020-04-30; First posted 2020-05-06 (Actual); Results first posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2021-08

CONDITIONS: Exocrine Pancreatic Insufficiency (EPI); Cystic Fibrosis (CF)
Keywords: Exocrine Pancreatic Insufficiency; EPI; Cystic Fibrosis; CF
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: 2, 2x2 Crossover
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MS1819 2240 mg/day vs PERT arm, (Active Comparator): Patients in arm will further be randomized to receive either the sequence consisting of MS1819 for 3 weeks followed by PERT for another 3 weeks or the opposite sequence of treatments, PERT for 3 weeks followed by MS1819 for another 3 weeks.
  Interventions: Drug: MS1819; Drug: Porcine PERT
- MS1819 4480 mg/day vs PERT arm (Active Comparator): Patients in arm will further be randomized to receive either the sequence consisting of MS1819 for 3 weeks followed by PERT for another 3 weeks or the opposite sequence of treatments, PERT for 3 weeks followed by MS1819 for another 3 weeks.
  Interventions: Drug: MS1819; Drug: Porcine PERT

INTERVENTIONS:
Drug: MS1819 — MS1819 in enteric capsules. It contains is a yeast-derived (non-porcine) lipase pancreatic enzyme replacement.
Drug: Porcine PERT — Porcine PERT is being used a comparator to MS1819 as a second drug/intervention.

SUMMARY:
The primary objectives of this study are to assess the safety and efficacy of MS1819 in enteric capsules vs porcine pancreatic enzyme replacement therapy (PERT) in patients with exocrine pancreatic insufficiency (EPI) due to cystic fibrosis (CF). The exploratory objective of the extension phase (EP) is to find a dose of MS1819 in immediate release capsules that is safe and results in CFA values in a therapeutic range.

DETAILED DESCRIPTION:
This is a Phase 2, open-label, multicenter, 2, 2x2 crossover study assessing the safety and efficacy of MS1819, 2240 mg/day vs porcine PERT, and 4480 mg/day vs porcine PERT given at the same dose and dosing regimen that was being administered during the pre-study period. MS1819 will be administered in enteric capsules.

MS1819 will be assessed in a 2x2 crossover including approximately 30 patients completing both periods. Fifteen patients will be randomized to the MS1819 2240 mg/day vs PERT arm, and 15 patients will be randomized to the MS1819 4480 mg/day vs PERT arm. Patients in each arm will further be randomized to receive either the sequence consisting of MS1819 for 3 weeks followed by PERT for another 3 weeks or the opposite sequence of treatments, PERT for 3 weeks followed by MS1819 for another 3 weeks.The coefficient of fat absorption (CFA) will be measured at the end of each 3 week study period. Patients enrolled into the extension phase (EP) will be composed of patients who have completed the crossover phase of OPTION 2.

ELIGIBILITY:
Inclusion Criteria:

1. Cystic fibrosis, based on 2 clinical features consistent with CF, plus either a new/historic sweat chloride ≥60 mmol/L (measured while not on a CFTR modulator) or genotype.
2. Under stable dose of porcine PERT
3. A fair or better nutritional status
4. Fecal elastase <100 µg/g
5. Standard-of-care medications including CFTR modulators are allowed

Exclusion Criteria:

1. History or diagnosis of fibrosing colonopathy
2. Any chronic diarrheal illness unrelated to pancreatic insufficiency
3. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥5 ×upper limit of normal (ULN), or total bilirubin level ≥1.5 ×ULN at the Screening visit
4. Feeding via an enteral tube during 6 months before screening
5. Forced expiratory volume ≤30% at the Screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (10):
  - Investigator Site 105, Long Beach, California
  - Investigator Site 102, Altamonte Springs, Florida
  - Investigator Site 107, Miami, Florida
  - Investigator Site 101, Glenview, Illinois
  - Investigator Site 111, Wichita, Kansas
  - Investigator Site 108, Portland, Maine
  - Investigator Site 103, Las Vegas, Nevada
  - Investigator Site 110, Cleveland, Ohio
  - Investigator Site 104, Toledo, Ohio
  - Investigator Site 106, Hershey, Pennsylvania
- Poland (5):
  - Investigator Site 205, Bialystok
  - Investigator Site 203, Karpacz
  - Investigator Site 206, Katowice
  - Investigator Site 202, Rabka-Zdrój
  - Investigator Site 204, Sopot

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients in extension arms only included patients who were already part of the initial phase of the study.
Groups:
- MS1819 (2240 mg/Day)-PERT Treatment Sequence: Patients were randomized to MS1819 (2240 mg/day) first and then PERT.
- PERT-MS1819 (2240 mg/Day) Sequence: Patients were randomized to PERT first and then MS1819 (2240 mg/day).
- MS1819 (4480 mg/Day)-PERT Treatment Sequence: Patients were first randomized to MS1819 (4480 mg/day) and then PERT.
- PERT-MS1819 (4480 mg/Day) Treatment Sequence: Patients were first randomized to PERT and then MS1819 (4480 mg/day)
- Extension MS1819 IR (4.4 g/Day): Regardless of previous treatment sequence in study patients received MS1819 IR 4.4 g/day
- Extension MS1819 (6.7 g/Day): Regardless of previous treatment sequence in study patients received MS1819 IR 6.7 g/day
Period: Crossover First and Second Interventions
Arm/Group | MS1819 (2240 mg/Day)-PERT Treatment Sequence | PERT-MS1819 (2240 mg/Day) Sequence | MS1819 (4480 mg/Day)-PERT Treatment Sequence | PERT-MS1819 (4480 mg/Day) Treatment Sequence | Extension MS1819 IR (4.4 g/Day) | Extension MS1819 (6.7 g/Day)
Started | 7 | 7 | 6 | 7 | 0 | 0
Completed | 6 | 6 | 5 | 7 | 0 | 0
Not Completed | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Period: Extension Phase
Arm/Group | MS1819 (2240 mg/Day)-PERT Treatment Sequence | PERT-MS1819 (2240 mg/Day) Sequence | MS1819 (4480 mg/Day)-PERT Treatment Sequence | PERT-MS1819 (4480 mg/Day) Treatment Sequence | Extension MS1819 IR (4.4 g/Day) | Extension MS1819 (6.7 g/Day)
Started | 0 (Only patients who completed period 1(Crossover: First and Second interventions) were eligible for participation in period 2.) | 0 (Only patients who completed period 1(Crossover: First and Second interventions) were eligible for participation in period 2.) | 0 (Only patients who completed period 1(Crossover: First and Second interventions) were eligible for participation in period 2.) | 0 (Only patients who completed period 1(Crossover: First and Second interventions) were eligible for participation in period 2.) | 9 (Although 24 participants were eligible for the Extension, not all elected to participate.) | 8 (Although 24 participants were eligible for the Extension, not all elected to participate.)
Completed | 0 | 0 | 0 | 0 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Modified intent to treat population.
Groups:
- Total: Total of all reporting groups
Arm/Group | MS1819 (2240 mg/Day)-PERT Treatment Sequence | PERT-MS1819 (2240 mg/Day) Sequence | MS1819 (4480 mg/Day)-PERT Treatment Sequence | PERT-MS1819 (4480 mg/Day) Treatment Sequence | Total
Number analyzed (Participants) | 6 | 7 | 5 | 7 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 5 | 7 | 25
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.2 (6.5) | 27.7 (4.1) | 27.4 (10.3) | 29.3 (4.3) | 27.3 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 4 | 12
  Male | 5 | 4 | 1 | 3 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 5 | 7 | 5 | 7 | 24
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety of MS1819 by Number of Subjects Reporting 1 or More Adverse Events
Description: Number of subjects reporting 1 or more adverse events
Time Frame: Each 3-week treatment period (crossover period) and 2-week treatment period (Extension period)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- MS1819 (2240 mg/Day): Patients were randomized to MS1819 (2240 mg/day) first and then PERT or PERT and then MS1819 (2240 mg/day)
- PERT ( MS1819 2240 mg/Day Crossover Group): Patients on PERT in MS1819 (2240 mg/day) - PERT or PERT-MS1819 (2240 mg/day) treatment sequences.
- MS1819 (4480 mg/Day): Patients were first randomized to MS1819 (4480 mg/day) and then PERT or or PERT and then MS1819 (4480 mg/day)
- PERT (MS1819 4480 mg/Day Crossover Group): Patients on PERT in MS1819 (4480 mg/day) - PERT or PERT-MS1819 (44800 mg/day) treatment sequences.
Arm/Group | MS1819 (2240 mg/Day) | PERT ( MS1819 2240 mg/Day Crossover Group) | MS1819 (4480 mg/Day) | PERT (MS1819 4480 mg/Day Crossover Group) | Extension MS1819 IR (4.4 g/Day) | Extension MS1819 (6.7 g/Day)
Number analyzed (Participants) | 14 | 13 | 13 | 12 | 9 | 8
Participants | 1 | 0 | 2 | 0 | 2 | 2

2. Primary Outcome: Efficacy of MS1819: Coefficient of Fat Absorption (CFA)
Description: The primary efficacy endpoint is the CFA that will be assessed at the end of each 3-week treatment period (crossover period) and 2-week treatment period (Extension period). CFAs for MS1819 will be compared to the CFAs of PERT using descriptive methods.
Time Frame: 6 weeks for crossover phase (to complete both first and second intervention) and 2 weeks for extension phase.
Population: Modified intent to treat
Measure: Mean (Standard Deviation); unit: percentage of fat absorption
Groups:
- MS1819 (2240 mg/Day): Patients on MS1819 in MS1819 (2240 mg/day) - PERT or PERT-MS1819 (2240 mg/day) treatment sequences.
- PERT (MS1819 2240 mg/Day Crossover Group): Patients on PERT in MS1819 (2240 mg/day) - PERT or PERT-MS1819 (2240 mg/day) treatment sequences.
- MS1819 (4480 mg/Day): Patients on MS1819 in MS1819 (4480 mg/day) - PERT or PERT-MS1819 (4480 mg/day) treatment sequences.
- PERT (MS1819 4480 mg/Day Crossover Group: Patients on PERT in MS1819 (4480 mg/day) - PERT or PERT-MS1819 (4480 mg/day) treatment sequences.
- Extension MS1819 IR (4.4 g/Day); Extension MS1819 IR (6.7g/Day): Patients enrolled in crossover phase
Arm/Group | MS1819 (2240 mg/Day) | PERT (MS1819 2240 mg/Day Crossover Group) | MS1819 (4480 mg/Day) | PERT (MS1819 4480 mg/Day Crossover Group | Extension MS1819 IR (4.4 g/Day) | Extension MS1819 IR (6.7g/Day)
Number analyzed (Participants) | 12 | 12 | 12 | 11 | 8 | 8
percentage of fat absorption | 66 (19.1) | 83.3 (13.1) | 52.8 (19.4) | 89.3 (4.7) | 52.9 (12.3) | 50.6 (9.2)

3. Secondary Outcome: Stool Weights
Description: The relative efficacy of MS1819 compared to porcine PERT will be assessed using stool weights.
Time Frame: Each 3-week treatment period (crossover period) and 2-week treatment period (Extension period)
Population: modified intent to treat
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | MS1819 (2240 mg/Day) | PERT (MS1819 2240 mg/Day Crossover Group) | MS1819 (4480 mg/Day) | PERT (MS1819 4480 mg/Day Crossover Group | Extension MS1819 IR (4.4 g/Day) | Extension MS1819 IR (6.7g/Day)
Number analyzed (Participants) | 12 | 12 | 12 | 11 | 8 | 8
grams | 1086.9 (609.2) | 664.4 (361.1) | 1689.6 (681.8) | 644.7 (310.1) | 1301.6 (478.7) | 1409.3 (448.0)

4. Secondary Outcome: Coefficient of Nitrogen Absorption (CNA)
Description: CNA that will be assessed at the end of each 3-week treatment period (crossover period) and 2-week treatment period (Extension period). CFAs for MS1819 will be compared to the CFAs of PERT using descriptive methods. CNAs for MS1819 will be compared to the CNAs of PERT using descriptive methods.
Time Frame: Each 3-week treatment period (crossover period) and 2-week treatment period (Extension period)
Population: modified intent to treat
Measure: Mean (Standard Deviation); unit: percentage of nitrogen absorption
Arm/Group | MS1819 (2240 mg/Day) | PERT (MS1819 2240 mg/Day Crossover Group) | MS1819 (4480 mg/Day) | PERT (MS1819 4480 mg/Day Crossover Group | Extension MS1819 IR (4.4 g/Day) | Extension MS1819 IR (6.7g/Day)
Number analyzed (Participants) | 12 | 12 | 12 | 11 | 8 | 8
percentage of nitrogen absorption | 94.4 (3.3) | 97.3 (1.8) | 90.9 (3.9) | 97.5 (1.0) | 93.1 (2.4) | 92.6 (2.5)

ADVERSE EVENTS:
Time Frame: Up to 15 weeks. The maximum overall duration for patients who participated in the crossover phase and extension phase, including screening and end of study visit was 15 weeks. The maximum overall duration for patients who participated in the crossover phase but did not participate in the extension phase, including screening and end of study visit was 11 weeks.
Arm/Group | MS1819 (2240 mg/Day) | PERT (MS1819 2240 mg/Day Crossover Group) | MS1819 (4480 mg/Day) | PERT (MS1819 4480 mg/Day Crossover Group | Extension MS1819 IR (4.4 g/Day) | Extension MS1819 IR (6.7g/Day)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13 | 0/13 | 0/12 | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/13 | 0/12 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 1/14 | 0/13 | 2/13 | 0/12 | 2/9 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MS1819 (2240 mg/Day) (N=14) | PERT (MS1819 2240 mg/Day Crossover Group) (N=13) | MS1819 (4480 mg/Day) (N=13) | PERT (MS1819 4480 mg/Day Crossover Group (N=12) | Extension MS1819 IR (4.4 g/Day) (N=9) | Extension MS1819 IR (6.7g/Day) (N=8)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/78/NCT04375878/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT04375878/SAP_001.pdf
  • Informed Consent Form (2020-04-23): https://cdn.clinicaltrials.gov/large-docs/78/NCT04375878/ICF_002.pdf